CLINICAL TRIAL: NCT00643578
Title: A Pilot Study to Evaluate the Dose-response of Inhaled Formoterol to Inhibit Airway Responsiveness to Methacholine in Patients With Mild Asthma
Brief Title: Dose-response of Inhaled Formoterol Using Methacholine Challenge as a Bioassay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Ivax-65307
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2011-11-18 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-11

CONDITIONS: Asthma
Keywords: formoterol; methacholine challenge
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Dry Powder Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): a single dose of 24 mcg of formoterol
  Interventions: Drug: formoterol; Device: Dry Powder Inhaler (Twisthaler)
- 1 (Active Comparator): a single dose of 12 mcg of formoterol
  Interventions: Drug: formoterol; Device: Dry Powder Inhaler (Twisthaler)

INTERVENTIONS:
Drug: formoterol — a single dose of 24 mcg of formoterol delivered by dry powder inhaler (Twisthaler)
  Arms: 2
Drug: formoterol — a single dose of 12 mcg of formoterol delivered by dry powder inhaler (Twisthaler)
  Arms: 1
Device: Dry Powder Inhaler (Twisthaler) — subjects inhaled deeply and forcefully and held their breath for 10 seconds for each dose

SUMMARY:
The purpose of this study is to find out whether a difference between two doses of formoterol can be detected by methacholine challenge.

DETAILED DESCRIPTION:
During the screening visit, subjects'vital signs (heart rate, blood pressure and temperature) will be measured and they will perform standard spirometry. If the results of this test are 70% of normal or greater, they will be examined by a physician, and blood (1 teaspoonful) and urine will be collected for routine laboratory tests (CBC and routine urinalysis). If they are a female, a pregnancy test will be performed.

During the second visit, subjects will inhale 1 or 2 doses of formoterol, (Foradil Aerolizer 12 mcg/capsule) a long-acting bronchodilator and 1 hour later, perform a methacholine test.

At the end of the methacholine test, they will be given albuterol to reverse the effects of methacholine. On the third study day, they will repeat the second visit but with the opposite dose of Foradil.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female 18 60 years of age, with a previous diagnosis of asthma that has been stable for at least 4 weeks and which is unlikely to exacerbate during the study because of, for example, seasonal allergen exposure. Women of childbearing age must not be pregnant or nursing, and must be using an acceptable method of contraception.
* Ability to perform ATS/ERS-acceptable and reproducible spirometry7
* Screening FEV1 ≥70% of predicted for height, age, sex, and race when short-acting inhaled bronchodilators are withheld for at least 6 hours
* At least a 20% decrease in FEV1 after inhaling ≤4 mg/mL of methacholine (i.e., a PC20 FEV1 ≤4 mg/mL)
* Can be taught to use the dry powder device in accordance with the product's medication guide.
* If using an oral inhaled or intranasal corticosteroid, dosage must be stable for at least 4 weeks.

Exclusion Criteria:

* Allergy or sensitivity to inhaled methacholine, formoterol or to other β2 agonists
* Intolerance to other components of the inhaler or sensitivity to milk proteins
* Cigarette smoking in past year or >10 pack-year smoking history
* Respiratory tract infection within the last four weeks
* History of severe asthma attack requiring hospitalization in the previous 12 months
* Short course of oral and/or systemic corticosteroids in the past 4 weeks
* Inability to withhold caffeinated beverages for 12 hours or medications for appropriate intervals prior to each methacholine challenge
* Require treatment with beta-blockers (administered by any route), MAO inhibitors, tricyclic antidepressants, and/or maintenance therapy with systemic corticosteroids
* History and/or presence of pulmonary conditions (including but not limited to cystic fibrosis and bronchiectasis) other than asthma
* History of clinically-significant cardiovascular, renal, neurologic, liver or endocrine dysfunction. Patients with well-controlled hypertension, hypercholesterolemia or diabetes will not be excluded.
* If female, a positive urine β-HCG test
* Known or suspected substance abuse (e.g., alcohol, marijuana, etc.) and/or any other medical or psychological conditions that in the investigator's opinion should preclude study enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hendeles, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Asthma Research Lab, Gainesville, Florida, United States

REFERENCES:
- [Background] Ahrens RC, Harris JB, Milavetz G, Annis L, Ries R. Use of bronchial provocation with histamine to compare the pharmacodynamics of inhaled albuterol and metaproterenol in patients with asthma. J Allergy Clin Immunol. 1987 Jun;79(6):876-82. doi: 10.1016/0091-6749(87)90235-1. PMID 3294976
- [Background] Blake KV, Hoppe M, Harman E, Hendeles L. Relative amount of albuterol delivered to lung receptors from a metered-dose inhaler and nebulizer solution. Bioassay by histamine bronchoprovocation. Chest. 1992 Feb;101(2):309-15. doi: 10.1378/chest.101.2.309. PMID 1310456
- [Background] Hendeles L, Beaty R, Ahrens R, Stevens G, Harman EM. Response to inhaled albuterol during nocturnal asthma. J Allergy Clin Immunol. 2004 Jun;113(6):1058-62. doi: 10.1016/j.jaci.2004.03.046. PMID 15208585
- [Background] Parameswaran KN, Inman MD, Ekholm BP, Morris MM, Summers E, O'Byrne PM, Hargreave FE. Protection against methacholine bronchoconstriction to assess relative potency of inhaled beta2-agonist. Am J Respir Crit Care Med. 1999 Jul;160(1):354-7. doi: 10.1164/ajrccm.160.1.9812035. PMID 10390425
- [Background] Ahrens RC, Hendeles L, Clarke WR, Dockhorn RJ, Hill MR, Vaughan LM, Lux C, Han SH. Therapeutic equivalence of Spiros dry powder inhaler and Ventolin metered dose inhaler. A bioassay using methacholine. Am J Respir Crit Care Med. 1999 Oct;160(4):1238-43. doi: 10.1164/ajrccm.160.4.9806101. PMID 10508813
- [Background] Creticos PS, Adams WP, Petty BG, Lewis LD, Singh GJ, Khattignavong AP, Molzon JA, Martinez MN, Lietman PS, Williams RL. A methacholine challenge dose-response study for development of a pharmacodynamic bioequivalence methodology for albuterol metered- dose inhalers. J Allergy Clin Immunol. 2002 Nov;110(5):713-20. doi: 10.1067/mai.2002.129036. PMID 12417879
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Background] Asmus MJ, Vaughan LM, Hill MR, Chesrown SE, Hendeles L. Stability of frozen methacholine solutions in unit-dose syringes for bronchoprovocation. Chest. 2002 May;121(5):1634-7. doi: 10.1378/chest.121.5.1634. PMID 12006455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April and November, 2008, the UF Asthma Research Lab recruited 37 patients for study.
Pre-assignment Details: Of the 37 subjects who signed informed consent, 25 did not meet inclusion/exclusion criteria. The provocational dose of methacholine causing a 20% drop in forced expiratory volume in the first second (PC20FEV1) was not less than or equal to 4 mg/mL.
Groups:
- Formoterol 12 First: a single dose of 12 mcg of formoterol was given first, then 24 mcg of formoterol
- Formoterol 24 First: a single dose of 24 mcg of formoterol was given first, then 12 mcg of formoterol
Period: Overall Study
Arm/Group | Formoterol 12 First | Formoterol 24 First
Started | 6 | 6
Completed | 4 | 6
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: A single dose of 12 mcg and 24 mcg, on separate days, of formoterol were given.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Post-dose PC20
Description: The PC20 is the provocational dose of methacholine causing a 20% drop in forced expiratory volume in the first second.
Time Frame: 3-7 days after visits 1 and 2
Population: Of the 12 subjects who qualified for randomization, 2 had a PC20 greater than 128 mg/mL (the maximum concentration of methacholine administered), after receiving 12 mcg of formoterol. Therefore, they were discontinued from the study since their PC20 would not be measurable with a higher dose of formoterol.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/mL
Groups:
- 12 Mcg Formoterol: low dose
- 24 Mcg Formoterol: high dose
Arm/Group | 12 Mcg Formoterol | 24 Mcg Formoterol
Number analyzed (Participants) | 10 | 10
mg/mL | 7 [2 to 22] | 16 [5 to 45]

2. Secondary Outcome: FEV1
Description: The forced expiratory volume in the first second, expressed as a percent predicted.
Time Frame: 1 hour after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent predicted
Groups:
- 12 Mcg of Formoterol: low dose
- 24 Mcg of Formoterol: high dose
Arm/Group | 12 Mcg of Formoterol | 24 Mcg of Formoterol
Number analyzed (Participants) | 10 | 10
percent predicted | 88 (12) | 91 (10)

ADVERSE EVENTS:
Groups:
- Formoterol 12: A single dose of 12 mcg of formoterol was administered.
- Formoterol 24: A single dose of 24 mcg of formoterol was administered.
Arm/Group | Formoterol 12 | Formoterol 24
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No